CLINICAL TRIAL: NCT05767463
Title: Correlation Between Pelvic Pain, Low Back Pain, and Postural Stability in Healthy Young Women During the Menstrual Cycle
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: October 6 University (Other)
Responsible Party: Principal Investigator, Hosam Magdy Metwally, Lecturer of physical therapy for neurology, October 6 University
Other Study IDs: 2023
Record Dates: First submitted 2023-03-01; First posted 2023-03-14 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Pain, Menstrual
Keywords: Pelvic pain, low back pain; Postural stability, and menstrual cycle
MeSH Terms: conditions — Dysmenorrhea; Pelvic Pain; Low Back Pain

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The menstrual cycle is governed by hormonal changes. Each cycle can be divided into three phases based on events in the ovary (ovarian cycle) or in the uterus (uterine cycle).

H0: There will be no correlation between pelvic pain and postural stability in healthy young women during the menstrual cycle H0: There will be no correlation between low back pain and postural stability in healthy young women during the menstrual cycle H0: There will be no correlation between pelvic pain and low back pain in healthy young women during the menstrual cycle

DETAILED DESCRIPTION:
Thirty-five female patients participated in this study. They were randomly assigned to the study. The outcome measures were pelvic pain assessed using the functional pelvic pain scale, low back pain assessed using the back pain functional scale, and postural stability assessed using the Biodex balance system.

ELIGIBILITY:
Inclusion Criteria:

1. All young females will suffer from pelvic pain, low back pain, and postural instability during the menstrual cycle
2. Age will range from 18 to 22 years
3. All young females will have a BMI range from 25-30

Exclusion Criteria:

1. Lumbar spondylosis
2. Lumbar disc prolapse
3. Sacroiliac joint arthritis
4. Low back trauma
5. BMI more than 30

Ages: 18 Years to 22 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: All young females will be recruited from the physical therapy faculty, October 6 University.
  All the assessment measurements will be done at the faculty of physical therapy, on October 6 University
Sampling Method: Probability Sample
Enrollment: 85 (Estimated)
Dates: Start 2022-11-22 (Actual); Primary Completion 2023-01-20 (Actual); Study Completion 2023-03-25 (Estimated)

PRIMARY OUTCOMES:
Functional pelvic pain scale | 30 days
  Functional Pelvic Pain Scale, designed to measure pelvic pain intensity as it relates to functions of daily living (bladder and bowel function, intercourse, walking, running, lifting, working, and sleeping),a total score is summed up out of 32. Furthermore, the maximum score obtained indicates the maximum physical disabilities of the patients. In addition, this scale also has an 'Adjusted score' ranging from 0 (0%)- no pain, normal function to 32 (100%)-cannot function because of pain.
Back pain functional scale | 30 days
  The Back Pain Functional Scale is a subjective scale used to measure the patient's physical function after low back pain. This scale was developed by Stratford et al. (2000), a total score is summed up out of 60. Furthermore, the maximum score obtained indicates the maximum physical abilities of the patients. In addition, this scale also has an 'Adjusted score' ranging from 0 (0%)-unable to perform any activity to 60 (100%)-no difficulty in any activity
Postural stability by using Biodex Balance System | 30 days
  The Biodex Balance System (BBS) has been used to evaluate postural balance. The BBS is a multiaxial device that objectively measures and records an individual's ability to stabilize the involved joint under dynamic stress

CONTACTS AND LOCATIONS:
Locations (1):
- October 6 University, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Undecided